CLINICAL TRIAL: NCT00948246
Title: EU Post-Market Study on Easyband®
Brief Title: European Union (EU) Post-Market Study on Easyband®
Status: Completed | Type: Observational
Sponsor: Allergan Medical (Industry)
Responsible Party: Sponsor
Organization: Allergan (Industry)
Other Study IDs: CIP10088
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2012-11-26 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2012-10

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Easyband: Subjects who had the Easyband device implanted laparoscopically.
  Interventions: Device: Easyband®

INTERVENTIONS:
Device: Easyband® — The Easyband adjustable gastric band device is implanted laparoscopically around the top of the stomach to create a small pouch. Adjustments to increase or decrease the stoma size are made non-invasively by telemetric connection between an internal and external antenna.

SUMMARY:
The purpose of this study is to collect additional safety, performance and effectiveness data of the Easyband gastric band medical device in the treatment of morbid obesity in 4 European countries where the device is a CE marked approved product.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrated failure in losing weight with non-invasive therapies
* BMI ≥ 40 kg/m2, or BMI ≥ 35 kg/m2 and < 40 kg/m2 with one or more significant medical conditions related to obesity

Exclusion Criteria:

* patients with BMI greater than 60 kg/m2
* patients who are not indicated for laparoscopic bariatric surgery
* patients with known allergies to implant materials such as silicone and PEEK
* patients whose abdominal structures have been damaged during preceding surgical procedures
* pregnant women
* patients under the age of 18 years
* patients treated with steroids
* patients addicted to alcohol or drugs, or who are mentally unstable, or who may not comply with the follow-up and dietary restrictions
* patients already implanted with a device sensitive to radio-frequency emissions such as implanted pacemaker, defibrillators, cochlear implants, implantable pumps etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Weight loss clinic and bariatric surgeon clinics within a hospital
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Brussels, Belgium
- Peschiera, Italy
- Nieuwegein, Netherlands
- Cheshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Easyband
Started | 110
Completed | 86
Not Completed | 24
Not completed — Lost to Follow-up | 11
Not completed — Adverse Event | 11
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Easyband
Number analyzed (Participants) | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 107
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 26
Region of Enrollment [Number; unit: participants]
  Belgium | 33
  Netherlands | 29
  Italy | 21
  United Kingdom | 27

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Ease of Implantation
Description: Percent of subjects whose device implantation was rated by the surgeon as a 1 or 2 on a 5-point scale, where 1 is "very easy" and 5 is "impossible."
Time Frame: < 1day
Population: Intent-to-treat
Measure: Number; unit: percentage of subjects
Arm/Group | Easyband
Number analyzed (Participants) | 110
percentage of subjects
  Introduction of Easyband into the abdomen | 71.8
  Placing Easyband around the stomach | 81.8
  Clipping of the Easyband around the stomach | 88.2

2. Secondary Outcome: % Excess Weight Loss
Description: Percent excess weight loss was defined as weight loss divided by excess weight multiplied by 100, where weight loss was equal to baseline weight minus follow-up weight, and excess weight was equal to baseline weight minus ideal weight.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: percentage of excess weight loss
Arm/Group | Easyband
Number analyzed (Participants) | 110
percentage of excess weight loss | 30.73 [29.389 to 35.128]

3. Secondary Outcome: Change in BMI
Description: Decrease in body mass index (BMI; measured in kg/m2) from baseline to 12 months
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: kg/m2
Arm/Group | Easyband
Number analyzed (Participants) | 110
kg/m2 | -7.23 [-7.898 to 6.560]

4. Secondary Outcome: Change in Weight
Description: Change in weight (in kilograms) at baseline to 12 months
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Easyband
Number analyzed (Participants) | 110
pounds | -20.70 [-22.754 to 18.640]

ADVERSE EVENTS:
Arm/Group | Easyband
Serious Adverse Events (participants affected / at risk) | 29/110
Other Adverse Events (participants affected / at risk) | 87/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Easyband (N=110)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Myocardial infarction (Cardiac disorders) | 1 (2)
Gastric dilatation (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Device malfunction (General disorders) | 3 (3)
Medical device complication (General disorders) | 5 (6)
Device related infection (Infections and infestations) | 1 (1)
Incision site infection (Infections and infestations) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Depression (Psychiatric disorders) | 2 (3)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1)
Medical device removal (Surgical and medical procedures) | 8 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Easyband (N=110)
Vomiting (Gastrointestinal disorders) | 42
Dysphagia (Gastrointestinal disorders) | 22
Abdominal pain upper (Gastrointestinal disorders) | 16
Constipation (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 8
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 6
Medical device complication (General disorders) | 9
Medical device pain (General disorders) | 7
Medical device removal (Surgical and medical procedures) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least one month prior to any proposed submission for publication or presentation of trial data, the PI will provide the Sponsor the manuscript for review, comment, and approval. No confidential information may be disclosed without Sponsor's written approval. If it is a multi-center trial, the first publication of the results shall be made in conjunction with the results from other Investigators at other centers.